CLINICAL TRIAL: NCT01209130
Title: An Open-Label, Multicenter, Phase I Trial of the Safety and Pharmacokinetics of Escalating Doses of DCDT2980S in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma and Chronic Lymphocytic Leukemia And DCDT2980S in Combination With Rituximab in Patients With Relapsed or Refractory B-Cell Non Hodgkin's Lymphoma
Brief Title: A Study of the Safety and Pharmacokinetics of Escalating Doses of DCDT2980S in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma and Chronic Lymphocytic Leukemia And DCDT2980S in Combination With Rituximab in Patients With Relapsed or Refractory B-Cell Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCT4862g; GO01295 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma, Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pinatuzumab vedotin; Rituximab

ARMS (2):
- A (Experimental)
  Interventions: Drug: DCDT2980S
- B (Experimental)
  Interventions: Drug: DCDT2980S; Drug: rituximab

INTERVENTIONS:
Drug: DCDT2980S — Intravenous repeating dose
Drug: rituximab — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase I, multicenter, open-label, dose-escalation study of DCDT2980S administered by intravenous (IV) infusion to patients with relapsed or refractory hematologic malignancies. In addition, at selected sites, DCDT2980S will be studied in combination with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* History of histologically-documented hematologic malignancy for which no effective standard therapy exists: indolent NHL (including Grades 1-3a FL; MZL [including splenic, nodal, and extra-nodal]; and SLL), Grade 3b FL, DLBCL, MCL, or CLL
* Must have at least one bi-dimensionally measurable lesion

Exclusion Criteria:

* Prior use of any monoclonal antibody or antibody-drug conjugate within 4 weeks prior to study treatment
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other investigational anti-cancer agent within 2 weeks prior to of study treatment
* Completion of autologous stem cell transplant within 100 days prior to study treatment
* Prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Throughout study or until early discontinuation

SECONDARY OUTCOMES:
Objective response, defined as a partial response (PR) or complete response (CR) | Throughout study or until early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (8):
- United States (8):
  - Stanford, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Hackensack, New Jersey
  - Portland, Oregon
  - Madison, Wisconsin